CLINICAL TRIAL: NCT01346410
Title: Phase IV Trial Evaluating the Use of Stereotactic Body Radiotherapy (SBRT) for the Treatment of Unresectable Pancreatic Cancer
Brief Title: Stereotactic Body Radiotherapy for Unresectable Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Kathy Baglan, MD, Radiation Oncologist, Mercy Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-060
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Stereotactic Radiation to Pancreas
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Suggested fractionation is 20-25 Gy / 1 fraction OR 30-36 Gy / 3 fractions (10-12 Gy per fraction) OR 40-45 Gy / 5 fractions (8-9 Gy per fraction)

SUMMARY:
This study will evaluate the local control rate as well as acute and late toxicity rates of stereotactic body radiotherapy (SBRT) for the treatment of unresectable pancreatic cancer.

DETAILED DESCRIPTION:
This is a single institution, non-randomized, prospective, phase IV trial of SBRT for unresectable pancreatic cancer.

Data collected will include patient demographics, pathology data, tumor stage, SBRT dose fractionation scheme, dose received by adjacent critical normal tissues, tumor recurrence data, and acute and late toxicities.

Follow up data will be collected during the patient's standard office visits. The anticipated duration of this study is 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >= 18 years
* Performance status of 0-3
* Unresectable pancreatic cancer
* Maximum tumor diameter < 7.5 cm
* Signed study-specific consent form

Exclusion Criteria:

* Maximum tumor diameter > 7.5 cm
* Prior radiotherapy to the upper abdomen
* Pregnant or lactating women, due to potential exposure of the fetus to RT and unknown effects of RT on lactating females
* Patients with psychiatric or addictive disorder that would preclude obtaining informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. John's Mercy Medical Center, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Radiation to Pancreas: Stereotactic Radiation to Pancreas
  Stereotactic Body Radiotherapy: Suggested fractionation is 20-25 Gy / 1 fraction OR 30-36 Gy / 3 fractions (10-12 Gy per fraction) OR 40-45 Gy / 5 fractions (8-9 Gy per fraction)
Period: Overall Study
Arm/Group | Stereotactic Radiation to Pancreas
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Radiation to Pancreas
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 79
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Local Control Rate
Description: Local recurrence is defined as tumor recurrence within the planning target volume. Local control rate will be evaluated by imaging techniques such as CT or MRI. Local recurrence will be defined as an increase of > 20% in tumor size. If necessary, a Positron Emission Tomography scan may be used to aid in diagnoses of local tumor recurrence.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiation to Pancreas
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Late Toxicity Rate
Description: Toxicities will be graded using CTCAE criteria at specified timepoints.
Time Frame: 5 years
Population: This outcome was not collected as planned.
Arm/Group | Stereotactic Radiation to Pancreas
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Stereotactic Radiation to Pancreas
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes